CLINICAL TRIAL: NCT06269510
Title: Enhancing Alcohol Treatment Engagement in ALD Patients
Brief Title: Enhancing Alcohol Treatment Engagement in Associated Liver Disease (ALD) Patients
Acronym: ENGAGE-ALD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jessica Mellinger, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17705; 1R01AA030748-01 (NIH)
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Alcohol-related Liver Disease; Liver Diseases
Keywords: Online web application; Engagement; Alcohol use disorder (AUD) treatment; Alcohol-related cirrhosis; SMART trial; Behavioral treatment
MeSH Terms: conditions — Liver Diseases; Alcoholism

STUDY DESIGN:
Intervention Model Description: Computer-generated urn randomization will ensure balanced groups based on stage of ALD (advanced ALD and non-advanced ALD) and inpatient versus outpatient status at time of recruitment. Second stage randomization to 3-month intervention conditions will be stratified based on response and non-response status. Urn randomization using stage of ALD and inpatient versus outpatient recruitment will also be used at the second stage randomization. Re-randomization of non-responders will be computerized and stratified by stage of ALD and inpatient vs outpatient status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Enhanced usual care (EUC) (Experimental): Eligible participants randomized will be given this for stage 1 of treatment (three months) and stage 2 (three months) if participants engaged in alcohol treatment during the first stage of treatment.
  Interventions: Behavioral: Enhanced Usual Care
- ENGAGE-ALD application (app) (Experimental): Eligible participants randomized to this arm will be given this for stage 1 (three months) of treatment and stage 2 (three months) if participants engaged in alcohol treatment during the first stage of treatment.
  Interventions: Behavioral: ENGAGE-ALD Application (APP)
- ENGAGE-ALD app then Treatment Facilitation Bundle (Experimental): Eligible participants randomized to this arm will be given this for stage 1 of treatment (three months). Participants that are non-responders (did not engage in alcohol treatment) will be re-randomized and assigned to the Treatment Facilitation bundle for stage 2 (three months).
  Interventions: Behavioral: ENGAGE-ALD Application (APP); Behavioral: Treatment Facilitation bundle
- Enhanced usual care then Treatment Facilitation Bundle (Experimental): Eligible participants randomized to this arm will be given this for stage 1 of treatment (three months). Participants that are non-responders (did not engage in alcohol treatment) will be re-randomized and assigned to the Treatment Facilitation bundle for stage 2 (three months).
  Interventions: Behavioral: Treatment Facilitation bundle; Behavioral: Enhanced Usual Care
- ENGAGE-ALD app then Enhanced usual care (Experimental): Eligible participants randomized to this arm will be given this for stage 1 (three months) of treatment. Participants that are non-responders (did not engage in alcohol treatment) will be re-randomized to the EUC arm stage 2 (three months).
  Interventions: Behavioral: ENGAGE-ALD Application (APP)
- Enhanced usual care then Enhanced usual care (Experimental): Eligible participants randomized to this arm will be given this for stage 1 of treatment (three months). Participants that are non-responders (did not engage in alcohol treatment) will be rerandomized to the Enhanced usual care arm stage 2 (three months).
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: ENGAGE-ALD Application (APP) — Participants randomized to this will complete the app at the time of enrollment.
  If in-person, will complete the app on a research laptop or iPad. The ENGAGE-ALD app consists of two modules developed based on preliminary data: 1) a misconception correction module and 2) a treatment matching module designed to match patients to participant's preferred form of alcohol treatment based on preferences for 19 different dimensions of alcohol treatment. The intervention will consist of administering a single session of the ENGAGE-ALD app.
  Arms: ENGAGE-ALD app then Enhanced usual care; ENGAGE-ALD app then Treatment Facilitation Bundle; ENGAGE-ALD application (app)
Behavioral: Treatment Facilitation bundle — Participants will complete a survey. The module includes motivational interviewing-informed content tailored to address and assist in overcoming barriers. After taking the survey, participants will receive a virtual coaching session (either via phone or online virtual platform). Sessions will focus on identifying participant goals with respect to alcohol use and liver health, providing education on risks of alcohol use to liver health and risks of relapse, reviewing participants individually identified barriers to alcohol treatment, exploring benefits of and these barriers to alcohol treatment, and performing collaborative goal-setting, among other topics.
  Arms: ENGAGE-ALD app then Treatment Facilitation Bundle; Enhanced usual care then Treatment Facilitation Bundle
Behavioral: Enhanced Usual Care — This group will receive standard hepatology care, and an educational pamphlet defining alcohol treatment resources available within Michigan Medicine and giving information on how participants can access these resources. This information will be given directly to participants that enroll in person or e-mailed to participants or sent via postal mail for those that enroll remotely.
  Arms: Enhanced usual care (EUC); Enhanced usual care then Enhanced usual care; Enhanced usual care then Treatment Facilitation Bundle

SUMMARY:
The purpose of this trial is to see if providing patients with alcohol-related liver disease with tailored alcohol use treatment options will increase engagement with treatment and correct possible misconceptions.

DETAILED DESCRIPTION:
Eligible participants will be randomized to stage 1 of treatment which consists of a previously pilot-tested behavioral application (app), the ENGAGE-ALD app, consisting of a knowledge improvement module and a preference-sensitive treatment matching module. Those who do not engage in AUD treatment after randomization ('non-responders') will be re-randomized at 3-months and continue on this in stage two if considered a responder (met treatment engagement). Participants that were not considered to have met "treatment engagement" will be re-randomized at 3-months to a Treatment Facilitation bundle consisting of a barriers to treatment survey followed by a health coaching session.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with all study procedures and availability for the duration of the study
* Willing and able to provide informed consent
* Enrolled at University of Michigan (UM) hepatology clinics or inpatients at UM Hospitals
* Documented diagnosis of alcohol-related liver disease (ALD) (per protocol)
* Recent alcohol use of any amount within the past 6 months as assessed by either patient interview, medical chart review, or positive alcohol biomarker (e.g. blood alcohol level, urinary ethyl glucuronide, urinary ethyl sulfate, or phosphatidylethanol) in the medical record.
* No alcohol use treatment within the past 1 month including, but not limited to:

  * Any professionally lead therapy with a mental health counselor (such as, one-on-one therapy, group therapy, couples or family therapy) with a primary aim of alcohol abstinence or reduction in alcohol use.
  * Community-based alcohol recovery groups (such as, Alcoholics Anonymous, SMART Recovery, Celebrate Recovery, Refuge Recovery)
  * Community-based church support groups primarily focused on alcohol abstinence or reduction in use.
  * Residential (inpatient) alcohol treatment
  * Intensive outpatient programs
  * Any telehealth version of the above options
* Access to a Smartphone or computer for purposes of follow-up. Those who do not have a Smartphone will be provided one along with a calling/data plan at no cost to subject by the study team for the duration of the research stud.
* Ability to speak and comprehend English

Exclusion Criteria:

* Unable to provide voluntary informed consent for any reason
* Substantially cognitively impaired as evidenced by Westhaven grade 2 or higher hepatic encephalopathy or a score >=10 on the Short Blessed Test for cognitive impairment.
* Unable to read or understand English
* Undergoing active evaluation for liver transplantation, is listed for liver transplant, or is post-transplantation
* Is enrolled in the multidisciplinary ALD clinic at Michigan Medicine
* Any other medical condition or circumstance that precludes safe and meaningful participation in the study
* History of nonadherence to previous clinical or research studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Alcohol treatment engagement | Baseline and six months
  Measured using self-report and defined as any single session (in-person or virtual) of the following:
  * Professional mental health counselor led one-on-one therapy, group therapy, couples, or family therapy with a primary aim of alcohol abstinence or reduction in alcohol use.
  * Community-based alcohol recovery groups (such as Alcoholics Anonymous, Self-Management and Recovery Training (SMART) Recovery, Celebrate Recovery, Refuge Recovery)
  * Community-based church support groups primarily focused on alcohol abstinence or reduction in use
  * Residential (inpatient) alcohol treatment
  * Intensive outpatient programs
  * Any telehealth version of the above options

SECONDARY OUTCOMES:
Alcohol Use Frequency as Measured by a 30-day alcohol recall calendar method | Baseline and six months
Percent heavy drinking days (PHDD) | Six months
  A heavy drinking day is defined as 5 or more drinks for men and 4 or more drinks for women.
Change in Liver health based on liver laboratory values (aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase) for all participants | Baseline and six months
Change in Liver health based on liver laboratory values (total bilirubin) for all participants | Baseline and six months
Change in Liver health based on The Model for End-Stage Liver Disease (MELD) score in participants with cirrhosis or alcoholic hepatitis | Baseline and six months
  Minimum MELD score: 6 points. Maximum MELD score: 40 points. Higher scores is considered a worse result.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Mellinger, MD, MSc, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No